CLINICAL TRIAL: NCT06112587
Title: Muscle Function and Strength Training of the Neck and Shoulder in Migraine and Tension-type Headache Patients.
Brief Title: Muscle Function and Strength Training of the Neck and Shoulder in Migraine and Tension-type Headache Patients. A Singel Arm Open Label Trial
Acronym: MUST-MITH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Bjarne Kjeldgaard Madsen, Principal Investigator, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHC F-23036562; Danish Headache center (Other: Rigshospitalet Glostrup)
Record Dates: First submitted 2023-10-10; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Migraine; Tension-Type Headache; Neck Pain
Keywords: migraine; tension-type headache; strength training; neck pain; exercise
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Neck Pain; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: A Single-Arm Open-Label Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Migraine and tension-type headache patients (Experimental): Patients diagnosed by a neurologist following the 3rd edition of the International Classification of Headaches Disorders (ICHD-III)
  Interventions: Behavioral: strength training

INTERVENTIONS:
Behavioral: strength training — A targeted 8-week strength-training course was offered as an intervention in combination with ergonomics and posture corrections and recommendations

SUMMARY:
A Single-Arm Open-Label Trial was performed at the Danish Headache Center (DHC), Department of Neurology, Rigshospitalet - Glostrup as part of the clinic.

Purpose:

To examine the effects of supervised group strength training and posture correction on headache frequency and muscle function around the neck and shoulders in patients with migraine and tension-type headaches.

Hypothesis:

Strength training of the neck and shoulders results in improved muscle function, which leads to a reduction in headache.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients with stable CGRP or botox.
* Tension type headache with no more than 5 migraine days/month.
* At least four days/months of headache at the moment of recruitment.

Exclusion Criteria:

* Pregnancy
* Post-traumatic headache, or headache that is likely to be associated with trauma.
* Significant psychiatric comorbidities, such as severe depression
* Medication Overuse Headaches.
* Severe arthrosis in the neck, shoulder, or disc herniation in the neck.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
headache frequency | two weeks prior to intervention, last two weeks of intervention
  number of days with headache

SECONDARY OUTCOMES:
neck pain maximal intensity | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  maximal neck pain intensity percieved by patient in a 0-10 NRPS
neck pain average intensity | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  average neck pain intensity percieved by patient in a 0-10 NRPS
neck pain frequency | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  number of days with neck pain
headache duration | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  hours with headache
medication intake | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  number of days with medication for pain taked
Functional level | Before intervention, after intervention and at 1 month follow up
  Self-reported limitated activities due to headache in a 0-10 scale thourgh the Patient-Specific Functional Scale
Headache average Intensity | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  average headache intensity percieved by patient in a 0-10 NRPS
Headache maximal Intensity | two weeks prior to intervention, last two weeks of intervention, and weeks 4 and 5 after intervention
  maximal headache intensity percieved by patient in a 0-10 NRPS
headache frequency | weeks 4 and 5 after intervention
  number of days with headache

OTHER OUTCOMES:
Maximal Voluntary Contraction of the Neck extension | Before intervention, after intervention and at 1 month follow up
  Maximal force of the neck extension (Newtons)
Maximal Voluntary Contraction of the Neck flexion | Before intervention, after intervention and at 1 month follow up
  Maximal force of the neck flexion (Newtons)
Maximal Voluntary Contraction of the Shoulder elevation | Before intervention, after intervention and at 1 month follow up
  Maximal force of the shoulder elevation (Newtons)
Moment arm for neck flexion and extension | Before intervention
  Distance between C7 and Protuberancia occipitalis (m)
Moment arm for shoulder elevation | Before intervention
  Distance between C7 and acromion of the right shoulder (m)
Moment arm for neck flexion | Before intervention, after intervention and at 1 month follow up
  Peak of the Maximal Voluntary Contraction x Moment arm of the neck flexion (N*m)
Moment arm of the neck extension | Before intervention, after intervention and at 1 month follow up
  Peak of the Maximal Voluntary Contraction x Moment arm of the neck extension (N*m)
Moment arm fof the shoulder elevation | Before intervention, after intervention and at 1 month follow up
  Peak of the Maximal Voluntary Contraction x Moment arm of the shoulder elevation (N*m)
Extension-Flexion ratio | Before intervention, after intervention and at 1 month follow up
  Ratio between moment arm of the neck extension and moment arm of the neck flexion.
Rate of force development of the shoulder elevation | Before intervention, after intervention and at 1 month follow up
  (75% of the peak value of the shoulder elevation (N) - 25% of the peak value of the shoulder elevation)/(time at de 75% of the peak of shoulder elevation (s) - time at 25% of the peak of shoulder elevation) in Newtons per second (N/s)
Early rate of force development of the shoulder elevation | Before intervention, after intervention and at 1 month follow up
  (Value of the peak of the shoulder elevation at 250ms after the 2,5% of the peak (N) - 2,5% of the peak value of the shoulder elevation)/0,250 (s) in Newtons per second (N/s)
Muscle tenderness | Before intervention, after intervention and at 1 month follow up
  Total Tenderness Score (0-48)
Muscle tenderness of the face | Before intervention, after intervention and at 1 month follow up
  Total Tenderness Score of the first 4 spots: masseter, coronoid process, temporalis and frontalis (0-24)
Muscle tenderness of the neck | Before intervention, after intervention and at 1 month follow up
  Total Tenderness Score of the last 4 spots: mastoid process, sternocleidmastoid, occipitalis and superior trapezius (0-24)
Craniocervical flexion score | Before intervention, after intervention and at 1 month follow up
  Craniocervical flexion test score. Possible values: 20, 22, 24, 26, 28 or 30 mmHg
Exercise sessions completed | During the intervention
  Number of training sessions performed by the participants
Percieved intensity | During the intervention
  Level of intensity percieved by patients in each exercise session
Intensity coherence | post-intervention
  Ratio between average of rate of percieved exertion by the patients and 10 (coefficient from 0 to 1).
Adherence of the programm | post-intervention
  Ratio between the number of exercise sessions completed by patients versus number of exercise sessions planned in the programm
Adherence to exercise | Week 1 to 5 after intervention
  Ratio between the number of exercise sessions completed after intervention until the follow-up.
Compliance of the programm | post-intervention
  Product between intensity coherence and adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: At the moment of publication and thereafter
Access Criteria: After its publication, according to the journal's policy and under the consensus of all authors.

REFERENCES:
- [Background] Steiner TJ, Gururaj G, Andree C, Katsarava Z, Ayzenberg I, Yu SY, Al Jumah M, Tekle-Haimanot R, Birbeck GL, Herekar A, Linde M, Mbewe E, Manandhar K, Risal A, Jensen R, Queiroz LP, Scher AI, Wang SJ, Stovner LJ. Diagnosis, prevalence estimation and burden measurement in population surveys of headache: presenting the HARDSHIP questionnaire. J Headache Pain. 2014 Jan 8;15(1):3. doi: 10.1186/1129-2377-15-3. PMID 24400999
- [Background] Linde M, Gustavsson A, Stovner LJ, Steiner TJ, Barre J, Katsarava Z, Lainez JM, Lampl C, Lanteri-Minet M, Rastenyte D, Ruiz de la Torre E, Tassorelli C, Andree C. The cost of headache disorders in Europe: the Eurolight project. Eur J Neurol. 2012 May;19(5):703-11. doi: 10.1111/j.1468-1331.2011.03612.x. Epub 2011 Dec 5. PMID 22136117
- [Background] Kroll LS, Callesen HE, Carlsen LN, Birkefoss K, Beier D, Christensen HW, Jensen M, Tomasdottir H, Wurtzen H, Host CV, Hansen JM. Manual joint mobilisation techniques, supervised physical activity, psychological treatment, acupuncture and patient education for patients with tension-type headache. A systematic review and meta-analysis. J Headache Pain. 2021 Aug 21;22(1):96. doi: 10.1186/s10194-021-01298-4. PMID 34418953
- [Background] Di Antonio S, Arendt-Nielsen L, Castaldo M. Cervical musculoskeletal impairments and pain sensitivity in migraine patients. Musculoskelet Sci Pract. 2023 Aug;66:102817. doi: 10.1016/j.msksp.2023.102817. Epub 2023 Jul 6. PMID 37451884
- [Background] Di Antonio S, Arendt-Nielsen L, Ponzano M, Bovis F, Torelli P, Pelosin E, Finocchi C, Castaldo M. Migraine patients with and without neck pain: Differences in clinical characteristics, sensitization, musculoskeletal impairments, and psychological burden. Musculoskelet Sci Pract. 2023 Aug;66:102800. doi: 10.1016/j.msksp.2023.102800. Epub 2023 Jun 14. PMID 37344290
- [Background] Ashina S, Bendtsen L, Lyngberg AC, Lipton RB, Hajiyeva N, Jensen R. Prevalence of neck pain in migraine and tension-type headache: a population study. Cephalalgia. 2015 Mar;35(3):211-9. doi: 10.1177/0333102414535110. Epub 2014 May 22. PMID 24853166
- [Background] Andersen LL, Suetta C, Andersen JL, Kjaer M, Sjogaard G. Increased proportion of megafibers in chronically painful muscles. Pain. 2008 Oct 31;139(3):588-593. doi: 10.1016/j.pain.2008.06.013. Epub 2008 Aug 12. PMID 18701218
- [Background] Madsen BK, Sogaard K, Andersen LL, Tornoe B, Jensen RH. Efficacy of strength training on tension-type headache: A randomised controlled study. Cephalalgia. 2018 May;38(6):1071-1080. doi: 10.1177/0333102417722521. Epub 2017 Jul 27. PMID 28750588
- [Background] Plotkin DL, Roberts MD, Haun CT, Schoenfeld BJ. Muscle Fiber Type Transitions with Exercise Training: Shifting Perspectives. Sports (Basel). 2021 Sep 10;9(9):127. doi: 10.3390/sports9090127. PMID 34564332
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Gago-Veiga AB, Camina Muniz J, Garcia-Azorin D, Gonzalez-Quintanilla V, Ordas CM, Torres-Ferrus M, Santos-Lasaosa S, Viguera-Romero J, Pozo-Rosich P. Headache: What to ask, how to examine, and which scales to use. Recommendations of the Spanish Society of Neurology's Headache Study Group. Neurologia (Engl Ed). 2022 Sep;37(7):564-574. doi: 10.1016/j.nrl.2018.12.006. Epub 2019 Mar 28. English, Spanish. PMID 30929913
- [Background] Madsen BK, Sogaard K, Andersen LL, Skotte JH, Jensen RH. Neck and shoulder muscle strength in patients with tension-type headache: A case-control study. Cephalalgia. 2016 Jan;36(1):29-36. doi: 10.1177/0333102415576726. Epub 2015 Apr 1. PMID 25834271
- [Background] Andersen LL, Nielsen PK, Sogaard K, Andersen CH, Skotte J, Sjogaard G. Torque-EMG-velocity relationship in female workers with chronic neck muscle pain. J Biomech. 2008;41(9):2029-35. doi: 10.1016/j.jbiomech.2008.03.016. Epub 2008 May 5. PMID 18460408
- [Background] Andersen LL, Andersen JL, Zebis MK, Aagaard P. Early and late rate of force development: differential adaptive responses to resistance training? Scand J Med Sci Sports. 2010 Feb;20(1):e162-9. doi: 10.1111/j.1600-0838.2009.00933.x. Epub 2009 May 26. PMID 19793220
- [Background] Maffiuletti NA, Aagaard P, Blazevich AJ, Folland J, Tillin N, Duchateau J. Rate of force development: physiological and methodological considerations. Eur J Appl Physiol. 2016 Jun;116(6):1091-116. doi: 10.1007/s00421-016-3346-6. Epub 2016 Mar 3. PMID 26941023
- [Background] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Background] Ashina H, Al-Khazali HM, Iljazi A, Ashina S, Amin FM, Schytz HW. Total tenderness score and pressure pain thresholds in persistent post-traumatic headache attributed to mild traumatic brain injury. J Headache Pain. 2022 Aug 8;23(1):96. doi: 10.1186/s10194-022-01457-1. PMID 35941545
- [Background] Bendtsen L, Jensen R, Jensen NK, Olesen J. Pressure-controlled palpation: a new technique which increases the reliability of manual palpation. Cephalalgia. 1995 Jun;15(3):205-10. doi: 10.1046/j.1468-2982.1995.015003205.x. PMID 7553810
- [Background] Horn KK, Jennings S, Richardson G, Vliet DV, Hefford C, Abbott JH. The patient-specific functional scale: psychometrics, clinimetrics, and application as a clinical outcome measure. J Orthop Sports Phys Ther. 2012 Jan;42(1):30-42. doi: 10.2519/jospt.2012.3727. Epub 2011 Oct 25. PMID 22031594
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Cummins D, Rivett DA, Thomas LC, Osmotherly PG. Reproduction and resolution of familiar head pain with upper cervical spine sustained joint mobilization may help identify cervicogenic headaches: a case-control study. J Man Manip Ther. 2023 Jun;31(3):198-205. doi: 10.1080/10669817.2022.2099181. Epub 2022 Jul 18. PMID 35844199
- [Background] Takasaki H, Yamasaki C. Immediate neck hypoalgesic effects of craniocervical flexion exercises and cervical retraction exercises among individuals with non-acute neck pain and a directional preference for retraction or extension: preliminary pretest-posttest randomized experimental design. J Man Manip Ther. 2023 Oct;31(5):368-375. doi: 10.1080/10669817.2023.2201918. Epub 2023 Apr 13. PMID 37052492
- [Background] van Ettekoven H, Lucas C. Efficacy of physiotherapy including a craniocervical training programme for tension-type headache; a randomized clinical trial. Cephalalgia. 2006 Aug;26(8):983-91. doi: 10.1111/j.1468-2982.2006.01163.x. PMID 16886935
- [Background] Andersen LL, Kjaer M, Andersen CH, Hansen PB, Zebis MK, Hansen K, Sjogaard G. Muscle activation during selected strength exercises in women with chronic neck muscle pain. Phys Ther. 2008 Jun;88(6):703-11. doi: 10.2522/ptj.20070304. Epub 2008 Mar 13. PMID 18339796
- [Background] Andersen LL, Kjaer M, Sogaard K, Hansen L, Kryger AI, Sjogaard G. Effect of two contrasting types of physical exercise on chronic neck muscle pain. Arthritis Rheum. 2008 Jan 15;59(1):84-91. doi: 10.1002/art.23256. PMID 18163419
- [Background] Fernandez-de-Las-Penas C, Cuadrado ML, Pareja JA. Myofascial trigger points, neck mobility, and forward head posture in episodic tension-type headache. Headache. 2007 May;47(5):662-72. doi: 10.1111/j.1526-4610.2006.00632.x. PMID 17501847
- [Background] Fernandez-de-Las-Penas C, Cuadrado ML, Pareja JA. Myofascial trigger points, neck mobility and forward head posture in unilateral migraine. Cephalalgia. 2006 Sep;26(9):1061-70. doi: 10.1111/j.1468-2982.2006.01162.x. PMID 16919056